CLINICAL TRIAL: NCT04246502
Title: A Phase 2,Randomized, Evaluate Efficacy and Safety of Capecitabine Plus Pyrotinib Versus Capecitabine Plus Trastuzumab and Pertuzumab in the First-line Treatment of HER2-positive Metastatic Breast Cancer
Brief Title: Capecitabine Plus Pyrotinib Versus Capecitabine Plus Trastuzumab and Pertuzumab in the First-line Treatment of HER2-positive Metastatic Breast Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shandong Cancer Hospital and Institute (Other)
Responsible Party: Principal Investigator, Zhiyong Yu, Shandong Breast Disease Centre, Shandong Cancer Hospital and Institute
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Shandong CHI-11
Record Dates: First submitted 2020-01-28; First posted 2020-01-29 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-01

CONDITIONS: Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Capecitabine; pyrotinib; Trastuzumab; pertuzumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A (Experimental)
  Interventions: Drug: Capecitabine and Pyrotinib
- B (Active Comparator)
  Interventions: Drug: Capecitabine,Trastuzumab, and Pertuzumab

INTERVENTIONS:
Drug: Capecitabine and Pyrotinib — Pyrotinib 400mg orally daily until progressive disease
  Arms: A
Drug: Capecitabine,Trastuzumab, and Pertuzumab — as instruction
  Arms: B

SUMMARY:
This is a randomized, multicenter phase 2 clinical trial to evaluate the efficacy and safety of capecitabine plus pyrotinib versus capecitabine plus trastuzumab plus pertuzumab in patients who have HER2 positive metastatic breast cancer and have not received systemic anticancer therapy for advanced disease.

ELIGIBILITY:
Inclusion Criteria:

* HER2 positive recurrent or metastasis breast cancer.
* Patients with measurable disease are eligible.
* Eastern Cooperative Oncology Group(ECOG) performance status 0 or 1.
* Adequate organ function.
* Signed, written inform consent obtained prior to any study procedure.

Exclusion Criteria:

* History of anti-cancer therapy for MBC（with the exception of one prior hormonal regimen for MBC）.
* History of HER tyrosine kinase inhibitors or monoclonal antibody for breast cancer in any treatment setting，except trastuzumab used in the neo-adjuvant or adjuvant setting.
* Assessed by the investigator to be unable receive systemic chemotherapy.
* History of other malignancy within the last 5 years，except for carcinoma in situ of cervix，basal cell carcinoma or squamous cell carcinoma of the skin that has been previously treated with curative intent.
* Pregnant or lactating women，or for women of childbearing potential unwilling to use a highly-effective contraception during of the study treatment and for at least 7 months after the last dose of study treatment.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2020-01 (Estimated); Primary Completion 2022-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival | Approximately 42 months

SECONDARY OUTCOMES:
Adverse Events and Serious Adverse Events | From the first drug administration to within 28 days for the last treatment
  AEs+SAEs
Overall Survival | Up to 2 years
Objective Response Rate | Approximately 42 months
Duration of Objective Response | Approximately 42 months
Clinical Benefit rate | From the start of randomization to 6 months